CLINICAL TRIAL: NCT04540289
Title: Personalised Risk scOre For Implantation of Defibrillators in Patients With Preserved LVEF>35% and a High Risk for Sudden Cardiac Death (PROFID-Preserved)
Brief Title: Personalised Risk scOre For Implantation of Defibrillators in Patients With Preserved LVEF>35% and a High Risk for Sudden Cardiac Death
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: trial is not feasible (very low event rates, no available risk predictor with acceptable predictive performance for discrimination of high-risk patients)
Sponsor: Helios Health Institute GmbH (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: LHI-2020-01; 847999 (Other Grant/Funding Number: European Union's Horizon 2020 research and innovation programme)
Record Dates: First submitted 2020-09-01; First posted 2020-09-07 (Actual); Last update posted 2023-03-08 (Actual); Status verified 2020-09

CONDITIONS: Myocardial Infarction; Sudden Cardiac Death
Keywords: Myocardial Infarction; Heart Failure; Sudden Cardiac Death; Implantable Cardioverter Defibrillator; PROFID; Personalized Medicine
MeSH Terms: conditions — Myocardial Infarction; Death, Sudden, Cardiac; Heart Failure | interventions — Defibrillators, Implantable

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The PROFID-Preserved trial is an open-label, blinded outcome assessment study. Thus, unblinding proce-dures for investigators are not applicable.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Optimal Medical Therapy without ICD device therapy (Active Comparator): Patients will be treated according to Optimal Medical Therapy defined by ESC Guidelines for treatment of patients with heart failure / chronic coronary syndromes and will not receive an ICD device
  Interventions: Drug: Optimal Medical Therapy (OMT)
- Optimal Medical Therapy with ICD device therapy (Experimental): Patients will be treated according to Optimal Medical Therapy defined by ESC Guidelines for treatment of patients with heart failure / chronic coronary syndromes and will receive an ICD device
  Interventions: Drug: Optimal Medical Therapy (OMT); Device: Implantable cardioverter-defibrillator (ICD)

INTERVENTIONS:
Drug: Optimal Medical Therapy (OMT) — Patients will be treated according to Optimal Medical Therapy defined by the following guidelines:
  1. 2019 ESC guidelines for the diagnosis and management of chronic coronary syndromes
  2. 2016 ESC guidelines for the management of acute and chronic heart failure
Device: Implantable cardioverter-defibrillator (ICD) — An ICD consists of an electronic medical device and electrode leads. The surgery can be performed in local anaesthesia, but a short general anaesthesia is required if the ICD has to be tested giving the patient an electric shock. Besides the possibility to shock during arrhythmias the ICD can potentially terminate ventricular tachycardias by rapid pacing for short periods (small bursts of pacing).
  The subcutaneous defibrillator is an established and valid alternative to the conventional ICD for the preven-tion of SCD. According to current guidelines, the subcutaneous defibrillator should be considered as an alternative to transvenous defibrillators in patients with an indication for an ICD when pacing therapy for bradycardia support, cardiac resynchronisation or antitachycardia pacing is not needed.
  Arms: Optimal Medical Therapy with ICD device therapy

SUMMARY:
The objective of the study is to demonstrate that in post-MI patients with preserved LVEF>35% but high risk for SCD according to a personalised risk score, the implantation of an ICD (index group) is superior to optimal medical therapy (control group) with respect to all-cause mortality.

DETAILED DESCRIPTION:
Sudden cardiac death (SCD) is a major public health problem, causing ~50% of cardiac fatalities and accounting for ~20% of all deaths in Europe. Identification of patients that are at risk for SCD and would benefit from ICD implantation is challenging. A predictor for increased risk of SCD after MI is a severely impaired heart function as expressed by a reduced left ventricular ejection fraction (LVEF). Based on this and on historical landmark trials, which found improved survival in patients with severely reduced LVEF who received an ICD, current clinical guidelines recommend prophylactic ICD implantation in post-MI patients with a LVEF ≤35% to improve overall survival by prevention of SCD. The current use of LVEF as sole patient stratification tool to guide treatment decisions for ICD implantation in patients with prior coronary event, as is currently recommended by clinical guidelines and performed in clinical practice, has significant limitations and results in substantial over- and undertreatment of patients. In particular, there is conclusive evidence that the majority of SCD cases occur in patients with only moderately reduced or preserved LVEF. Thus, with current guidelines most of patients that will develop SCD are not protected by means of ICD implantation.

The objective of the study is to demonstrate that in post-MI patients with preserved LVEF>35% but high risk for SCD according to a personalised risk score, the implanta-tion of an ICD (index group) is superior to optimal medical therapy (control group) with respect to all-cause mortality.

PROFID-Preserved is a non-commercial, investigator-driven, prospective, parallel-group, randomised, open-label, blinded outcome assessment (PROBE), multi-centre, superiority trial without dedicated investigational medical device (Proof of Strategy Trial) with two groups with 1:1 randomi-sation. It will be conducted in about 12 European countries with more than 150 clinical sites participating.

This study is an event driven trial and the number of randomised patients is estimated to be 1,440, required to collect 297 first primary outcome events within 30 months of mean follow-up.

Total study duration:

Enrolment of 30 months. All patients will be followed until 297 valid primary endpoints are reached (event-driven trial) which is expected about 15 months after last patient in. Total study duration of 47 months is expected which might be adapted based on a blinded interim analysis of the overall occurrence of the primary endpoint.

Individual study duration:

Expected median follow-up time will be about 30 months per patient with a minimum follow-up time of 15 months and a maximum follow-up time of presumably 45 months.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years.
* Documented history of myocardial infarction either as ST segment elevation myocardial infarction (STEMI) or as non-ST segment elevation myocardial infarction (NSTEMI).
* LVEF > 35% at transthoracic echocardiography or cardiac magnetic resonance imaging (MRI).
* Predicted personalised annual risk of SCD according to the clinical risk calculator >3%.
* Signed informed consent.

Exclusion Criteria:

* Class I or IIa indication for implantation of an ICD for secondary prevention of sudden cardiac death and ventricular tachycardia (according to the 2015 ESC Guidelines for the management of patients with ventricular arrhythmias and the prevention of sudden cardiac death, see Appendix V).
* Ventricular tachycardia induced in an electrophysiologic study.
* Unexplained syncope when ventricular arrhythmia is suspected as the cause of syncope.
* Conclusive clinical indication for CRT (class I or IIa indication according to the 2016 ESC Guidelines for the diagnosis and treatment of acute and chronic heart failure)
* Carrying any implanted cardiac pacemaker, defibrillator or CRT device.
* Violation of instruction for use (IFU) of the selected ICD device by at least one of the random group treatments.
* Hospitalised with unstable heart failure with NYHA class IV within 1 month prior to enrolment.
* Acute coronary syndrome or cardiac revascularization therapy by coronary angioplasty or coronary artery bypass grafting within 3 months prior to enrolment.
* Cardiac valve surgery or percutaneous cardiac valvular intervention such as transcatheter aortic valve replacement or transcatheter mitral valve repair performed within 3 months prior to enrolment.
* On the waiting list for heart transplantation.
* Any known disease that limits life expectancy to less than 1 year.
* Participation in another clinical trial, either within the 3 months prior to enrolment or still on-going (participation in sub-studies connected to this trial is permitted).
* Previous participation in PROFID-Preserved.
* Drug abuse or clinically manifest alcohol abuse.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2023-01-31 (Actual); Study Completion 2023-01-31 (Actual)

PRIMARY OUTCOMES:
Time from randomisation to the occurrence of all-cause death | Randomization to end of study (event-driven, expected about 15 months after last patient in)

SECONDARY OUTCOMES:
Time from randomisation to death from cardivascular causes | Randomization to end of study (event-driven, expected about 15 months after last patient in)
Time from randomisation to sudden cardiac death | Randomization to end of study (event-driven, expected about 15 months after last patient in)
Time from randomisation to first hospital readmissions for cardiovascular causes after randomisation | Randomization to end of study (event-driven, expected about 15 months after last patient in)
Average length of stay in hospital during the study period | Randomization to end of study (event-driven, expected about 15 months after last patient in)
Quality of life (EQ-5D-5L) trajectories over time | At baseline and 6-month intervals thereafter

CONTACTS AND LOCATIONS:
Overall Officials: Gerhard Hindricks, MD, Principal Investigator — Department of Electrophysiology, Leipzig Heart Center at University of Leipzig; Nikolaos Dagres, MD, Principal Investigator — Department of Electrophysiology, Leipzig Heart Center at University of Leipzig

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Related Info — https://profid-project.eu/